CLINICAL TRIAL: NCT02684851
Title: The Use of Tranexamic Acid to Reduce Blood Loss in Acetabular Surgery
Acronym: TXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-12-06B
Record Dates: First submitted 2016-02-11; First posted 2016-02-18 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-01

CONDITIONS: Acetabular Fractures
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Inactive
  Interventions: Drug: Placebo
- Tranexamic (Active Comparator): Tranexamic acid: anti-fibrinolytic agents
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid: anti-fibrinolytic agents
  Other Names: Tranexamic acid (anti-fibrinolytic agents )
  Arms: Tranexamic
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if patients undergoing acetabular ORIF (open reduction with internal fixation) who receive tranexamic acid have a reduced risk of allogenic blood transfusion, perioperative blood loss, wound complication and higher risk for thromboembolic events compared to patients who receive placebo. Investigators want to determine the cost-effectiveness related to allogenic blood transfusion as a blood loss management strategy in acetabular open reduction internal fixation (ORIF). Orthopaedic surgery carries with it a significant risk for blood loss. Current management of perioperative blood loss is the use of allogenic blood transfusion. Allogenic blood transfusion carries with it a risk for HIV and Hepatitis C as well as multiple adverse reactions. There have been significant efforts to reduce the use of allogenic blood transfusion in orthopaedic surgery. Tranexamic acid, an anti-fibrinolytic agent, has been used in management of blood during surgery. In order to determine the impact of tranexamic acid in reducing blood loss among patients undergoing acetabular ORIF, investigators will conduct a prospective randomized study. Patients undergoing acetabular surgery will be screened for this study. Patients will be then randomized to placebo or tranexamic acid which will be administered during and after surgery. The following data will be collected: patient characteristics, surgery information, blood loss, blood transfusions, wound complication within 30 days of surgery, and cost.

DETAILED DESCRIPTION:
In this study, investigators plan to prospectively determine the effect of tranexamic acid on blood loss and outcome after surgery to the acetabulum.

Patients will be randomized into two groups. In this study, investigators plan to administer a 10mg/kg dose within 30 minutes of surgery followed by a 10mg/kg infusion over a 4hr period to the treatment group (for patients weighting over 100kg, a weight of 100kg will be used for the dose calculation). The control group will receive equal volumes of and rates of normal saline.

Research Questions:

1. Do patients undergoing acetabular ORIF who receive tranexamic acid have a reduced risk of allogenic blood transfusion as compared to patients who receive placebo?
2. Do patients undergoing acetabular ORIF who receive tranexamic acid have reduced peri-operative blood loss as compared to patients who receive placebo?
3. Do patients undergoing acetabular ORIF who receive tranexamic acid have a higher risk for thromboembolic events than patients who receive placebo?
4. Do patients undergoing acetabular ORIF who receive tranexamic acid have a reduced risk of wound complications (prolonged wound drainage, return to the OR within 30 days, infection)?
5. Is the use of tranexamic acid cost effective relative to the use of allogenic blood transfusion as a blood loss management strategy in acetabular ORIF?

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or above undergoing acetabular ORIF.

Exclusion Criteria:

* All patients aged below 18 years undergoing acetabulum surgery
* Patients with color-blindness (color vision changes used to assess toxicity)
* Patients with subarachnoid hemorrhage.
* Patients with active intravascular coagulation.
* Patients with a previous history of venous thromboembolism or with a history of hypercoaguable conditions (i.e. Factor V Leiden, antiphospholipid antibody).
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-10; Primary Completion 2016-07-25 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Karunakar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - University of Missouri, Columbia, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Astedt B, Liedholm P, Wingerup L. The effect of tranexamic acid on the fibrinolytic activity of vein walls. Ann Chir Gynaecol. 1978;67(6):203-5. PMID 742821
- [Background] Benoni G, Fredin H, Knebel R, Nilsson P. Blood conservation with tranexamic acid in total hip arthroplasty: a randomized, double-blind study in 40 primary operations. Acta Orthop Scand. 2001 Oct;72(5):442-8. doi: 10.1080/000164701753532754. PMID 11728069
- [Background] Benoni G, Lethagen S, Fredin H. The effect of tranexamic acid on local and plasma fibrinolysis during total knee arthroplasty. Thromb Res. 1997 Feb 1;85(3):195-206. doi: 10.1016/s0049-3848(97)00004-2. PMID 9058494
- [Background] Benoni G, Lethagen S, Nilsson P, Fredin H. Tranexamic acid, given at the end of the operation, does not reduce postoperative blood loss in hip arthroplasty. Acta Orthop Scand. 2000 Jun;71(3):250-4. doi: 10.1080/000164700317411834. PMID 10919295
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Callaghan JJ, Spitzer AI. Blood management and patient specific transfusion options in total joint replacement surgery. Iowa Orthop J. 2000;20:36-45. PMID 10934623
- [Background] Carson JL, Altman DG, Duff A, Noveck H, Weinstein MP, Sonnenberg FA, Hudson JI, Provenzano G. Risk of bacterial infection associated with allogeneic blood transfusion among patients undergoing hip fracture repair. Transfusion. 1999 Jul;39(7):694-700. doi: 10.1046/j.1537-2995.1999.39070694.x. PMID 10413276
- [Background] Claeys MA, Vermeersch N, Haentjens P. Reduction of blood loss with tranexamic acid in primary total hip replacement surgery. Acta Chir Belg. 2007 Jul-Aug;107(4):397-401. doi: 10.1080/00015458.2007.11680081. PMID 17966532
- [Background] Clark CR. Perioperative blood management in total hip arthroplasty. Instr Course Lect. 2009;58:167-72. PMID 19385529
- [Background] Eikelboom JW, Karthikeyan G, Fagel N, Hirsh J. American Association of Orthopedic Surgeons and American College of Chest Physicians guidelines for venous thromboembolism prevention in hip and knee arthroplasty differ: what are the implications for clinicians and patients? Chest. 2009 Feb;135(2):513-520. doi: 10.1378/chest.08-2655. PMID 19201714
- [Background] Ekback G, Axelsson K, Ryttberg L, Edlund B, Kjellberg J, Weckstrom J, Carlsson O, Schott U. Tranexamic acid reduces blood loss in total hip replacement surgery. Anesth Analg. 2000 Nov;91(5):1124-30. doi: 10.1097/00000539-200011000-00014. PMID 11049894
- [Background] Fergusson DA, Hebert PC, Mazer CD, Fremes S, MacAdams C, Murkin JM, Teoh K, Duke PC, Arellano R, Blajchman MA, Bussieres JS, Cote D, Karski J, Martineau R, Robblee JA, Rodger M, Wells G, Clinch J, Pretorius R; BART Investigators. A comparison of aprotinin and lysine analogues in high-risk cardiac surgery. N Engl J Med. 2008 May 29;358(22):2319-31. doi: 10.1056/NEJMoa0802395. Epub 2008 May 14. PMID 18480196
- [Background] Garneti N, Field J. Bone bleeding during total hip arthroplasty after administration of tranexamic acid. J Arthroplasty. 2004 Jun;19(4):488-92. doi: 10.1016/j.arth.2003.12.073. PMID 15188109
- [Background] Gill JB, Rosenstein A. The use of antifibrinolytic agents in total hip arthroplasty: a meta-analysis. J Arthroplasty. 2006 Sep;21(6):869-73. doi: 10.1016/j.arth.2005.09.009. PMID 16950041
- [Background] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586
- [Background] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Background] Haynes RB, et al. Clinical Epidemiology: How to Do Clinical Practice Research. 3rd ed. Lippincott Williams and Wilkins, 2006.
- [Background] Husted H, Blond L, Sonne-Holm S, Holm G, Jacobsen TW, Gebuhr P. Tranexamic acid reduces blood loss and blood transfusions in primary total hip arthroplasty: a prospective randomized double-blind study in 40 patients. Acta Orthop Scand. 2003 Dec;74(6):665-9. doi: 10.1080/00016470310018171. PMID 14763696
- [Background] Ido K, Neo M, Asada Y, Kondo K, Morita T, Sakamoto T, Hayashi R, Kuriyama S. Reduction of blood loss using tranexamic acid in total knee and hip arthroplasties. Arch Orthop Trauma Surg. 2000;120(9):518-20. doi: 10.1007/s004029900132. PMID 11011672
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Karunakar MA, Shah SN, Jerabek S. Body mass index as a predictor of complications after operative treatment of acetabular fractures. J Bone Joint Surg Am. 2005 Jul;87(7):1498-502. doi: 10.2106/JBJS.D.02258. PMID 15995116
- [Background] Klein HG, Spahn DR, Carson JL. Red blood cell transfusion in clinical practice. Lancet. 2007 Aug 4;370(9585):415-26. doi: 10.1016/S0140-6736(07)61197-0. PMID 17679019
- [Background] Munoz M, Garcia-Erce JA, Villar I, Thomas D. Blood conservation strategies in major orthopaedic surgery: efficacy, safety and European regulations. Vox Sang. 2009 Jan;96(1):1-13. doi: 10.1111/j.1423-0410.2008.01108.x. PMID 19121192
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Niskanen RO, Korkala OL. Tranexamic acid reduces blood loss in cemented hip arthroplasty: a randomized, double-blind study of 39 patients with osteoarthritis. Acta Orthop. 2005 Dec;76(6):829-32. doi: 10.1080/17453670510045444. PMID 16470437
- [Background] Orpen NM, Little C, Walker G, Crawfurd EJ. Tranexamic acid reduces early post-operative blood loss after total knee arthroplasty: a prospective randomised controlled trial of 29 patients. Knee. 2006 Mar;13(2):106-10. doi: 10.1016/j.knee.2005.11.001. Epub 2006 Feb 17. PMID 16487712
- [Background] Rajesparan K, Biant LC, Ahmad M, Field RE. The effect of an intravenous bolus of tranexamic acid on blood loss in total hip replacement. J Bone Joint Surg Br. 2009 Jun;91(6):776-83. doi: 10.1302/0301-620X.91B6.22393. PMID 19483232
- [Background] Rosencher N, Kerkkamp HE, Macheras G, Munuera LM, Menichella G, Barton DM, Cremers S, Abraham IL; OSTHEO Investigation. Orthopedic Surgery Transfusion Hemoglobin European Overview (OSTHEO) study: blood management in elective knee and hip arthroplasty in Europe. Transfusion. 2003 Apr;43(4):459-69. doi: 10.1046/j.1537-2995.2003.00348.x. PMID 12662278
- [Background] Sadeghi M, Mehr-Aein A. Does a single bolus dose of tranexamic acid reduce blood loss and transfusion requirements during hip fracture surgery? A prospective randomized double blind study in 67 patients. Acta Medica Iranica 2007; 45: 437-42.
- [Background] Salido JA, Marin LA, Gomez LA, Zorrilla P, Martinez C. Preoperative hemoglobin levels and the need for transfusion after prosthetic hip and knee surgery: analysis of predictive factors. J Bone Joint Surg Am. 2002 Feb;84(2):216-20. doi: 10.2106/00004623-200202000-00008. PMID 11861727
- [Background] Scannell BP, Loeffler BJ, Bosse MJ, Kellam JF, Sims SH. Efficacy of intraoperative red blood cell salvage and autotransfusion in the treatment of acetabular fractures. J Orthop Trauma. 2009 May-Jun;23(5):340-5. doi: 10.1097/BOT.0b013e31819f691d. PMID 19390361
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Stulberg BN, Zadzilka JD. Blood management issues using blood management strategies. J Arthroplasty. 2007 Jun;22(4 Suppl 1):95-8. doi: 10.1016/j.arth.2007.03.002. PMID 17570287
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Tornetta P 3rd. Displaced acetabular fractures: indications for operative and nonoperative management. J Am Acad Orthop Surg. 2001 Jan-Feb;9(1):18-28. doi: 10.5435/00124635-200101000-00003. PMID 11174160
- [Background] Westrich GH, Bottner F, Windsor RE, Laskin RS, Haas SB, Sculco TP. VenaFlow plus Lovenox vs VenaFlow plus aspirin for thromboembolic disease prophylaxis in total knee arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):139-43. doi: 10.1016/j.arth.2006.05.017. PMID 16950076
- [Background] Westrich GH, Sculco TP. Prophylaxis against deep venous thrombosis after total knee arthroplasty. Pneumatic plantar compression and aspirin compared with aspirin alone. J Bone Joint Surg Am. 1996 Jun;78(6):826-34. doi: 10.2106/00004623-199606000-00004. PMID 8666599
- [Background] Zufferey P, Merquiol F, Laporte S, Decousus H, Mismetti P, Auboyer C, Samama CM, Molliex S. Do antifibrinolytics reduce allogeneic blood transfusion in orthopedic surgery? Anesthesiology. 2006 Nov;105(5):1034-46. doi: 10.1097/00000542-200611000-00026. PMID 17065899
- [Background] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tranexamic
Started | 42 | 45
Completed | 42 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tranexamic | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Customized [Mean (Standard Deviation); unit: Years] | 43.7 (13.5) | 42.3 (16.2) | 43.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 32 | 32 | 64
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (13.5) | 32.1 (16.2) | 31.7 (14.7)
Co-morbidities [Count of Participants; unit: Participants]
  Cardiac Disease | 2 | 1 | 3
  Diabetes | 5 | 5 | 10
Surgical approach [Count of Participants; unit: Participants]
  Posterior Approach | 37 | 35 | 72
  Anterior Approach | 4 | 6 | 10
  Combined Anterior/Posterior | 1 | 4 | 5
Operative time in minutes [Mean (Standard Deviation); unit: Minutes] | 239.4 (100.6) | 209.9 (72.3) | 224.7 (86.6)
Preoperative Hemoglobin in g/dl [Mean (Standard Deviation); unit: g/dl] | 11.1 (2.26) | 11.9 (2.19) | 11.5 (2.23)
Letournel Fracture Classification [Count of Participants; unit: Participants] — Elementary Type include posterior wall, posterior column, anterior column, anterior wall and transverse acetabular fractures.
  Associated type include transverse posterior wall, posterior column/posterior wall, anterior column posterior hemitranscerse, t-type and associated both column acetabular fractures.
  Participants
    Associated Fractures | 22 | 17 | 39
    Elementary Fractures | 20 | 28 | 48
Orthopaedic Trauma Association Fracture Classification [Count of Participants; unit: Participants]
  Pelvis, acetabulum, partial articular, isolated column and/or wall fracture (62A) | 22 | 28 | 50
  Pelvis, acetabulum, partial articular, transverse type fracture (62B) | 14 | 13 | 27
  Pelvis, acetabulum, complete articular, associated both column fracture (62C) | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Allogenic Blood Transfusion Rates
Description: Number of participant received allogenic blood transfusions.
Time Frame: post-operative
Measure: Count of Participants; unit: Participants
Groups:
- Tranexamic: Patients in the intervention group were administered a 10mg/kg preoperative dose of tranexamic acid within 30 minutes prior to surgery followed by a 10mg/kg infusion over a 4hr period during surgery (for patients weighing over 100kg, a weight of 100kg was used for the dose calculation).
- Placebo: Patients in the control group received an equal volume and rate of normal saline. Patients and providers were blinded with the aid of an investigational drug pharmacy.
Arm/Group | Tranexamic | Placebo
Number analyzed (Participants) | 45 | 42
Participants | 21 | 13

2. Primary Outcome: Units of Packed Red Blood Cells Transfused
Description: Average units packed red blood cells transfused among participants
Time Frame: perioperative
Measure: Mean (Standard Deviation); unit: Units of packed red blood cells
Arm/Group | Tranexamic | Placebo
Number analyzed (Participants) | 45 | 42
Units of packed red blood cells | 2.65 (1.27) | 2.36 (0.81)

3. Secondary Outcome: Number of Participants With a Thromboembolic Event
Description: Do patients undergoing acetabular ORIF who receive tranexamic acid have a higher risk for thromboembolic events than patients who receive placebo?
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic | Placebo
Number analyzed (Participants) | 45 | 42
Participants | 1 | 0

4. Secondary Outcome: Estimate Blood Loss
Description: To measure average estimate perioperative blood loss
Time Frame: perioperative
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic | Placebo
Number analyzed (Participants) | 45 | 42
mL | 727.6 (702.52) | 560.1 (378.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tranexamic | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/42
Other Adverse Events (participants affected / at risk) | 0/45 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic (N=45) | Placebo (N=42)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-04-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02684851/Prot_SAP_000.pdf
  • Informed Consent Form (2013-04-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02684851/ICF_001.pdf